CLINICAL TRIAL: NCT06220305
Title: DNA Methylation Combined With Artificial Intelligence Imaging for Early Benign and Malignant Differentiation of Lung Nodules:an Observational,Single-center Clinical Trial(MAGIC Study)
Brief Title: DNA Methylation Combined With Artificial Intelligence Imaging to Identify Lung Nodules
Acronym: MAGIC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 2023SR257
Record Dates: First submitted 2024-01-14; First posted 2024-01-23 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Lung Cancer Diagnosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pulmonary Nodule Group: patient conform pulmonary nodules on CT images
  Interventions: Diagnostic Test: DNA methylation joint AI imaging

INTERVENTIONS:
Diagnostic Test: DNA methylation joint AI imaging — DNA were extracted from patients'plasma ,then the DNA was bisulfite converted and tested by DNA methylation assay.The results were combined with AI images to differentiate between benign and malignant lung nodules.

SUMMARY:
Lung cancer is the leading cause of cancer deaths,and the key to reducing mortality in lung cancer patients is early diagnosis and treatment.Currently,peripheral blood DNA methylation is a novel in vitro molecular marker for tumors.Meanwhile artificial intelligence diagnostic system can further improve the diagnostic ability.The purpose of this study is to apply the overall DNA methylation level (i.e.,methylation profile) and the altered methylation degree of specific genes as tumor diagnostic indexes,and combined with the artificial intelligence imaging technology for the early and accurate diagnosis of lung cancer,to achieve the early detection,diagnosis,and treatment of lung cancer,and to effectively reduce the mortality rate of lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* (1) Patients with pulmonary nodules diagnosed by imaging;
* (2) No contraindications to blood collection;
* (3) Voluntary completed DNA methylation testing;
* (4) Signed informed consent and performed all the study mandated procedures.

Exclusion Criteria:

* (1) Pregnant or lactating(6 months) women;
* (2) History of malignancy or known malignancy or precancerous lesions or known tuberculosis within 3 years;
* (3) Autoimmune system disorders;
* (4) Undergoing any diagnostic puncture therapy, such as percutaneous lung biopsy, transbronchial, pre-enrollment biopsy, or surgical procedures (within 6 months); (5) Recipients of organ transplants or prior non-autologous (allogeneic) bone marrow transplants or stem cell transplants; (6) Received antibiotic therapy within 14 days or applied a drug that elevates white blood cells within 45 days prior to the blood draw.

Ages: 20 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with single pulmonary nodule found by CT scan.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy of early diagnosis of benign and malignant lung nodules by blood DNA methylation results combined with AI imaging | 10 months
  Construction of a diagnostic model for DNA methylation combined with AI imaging. Comparing the results of the model with pathologic diagnosis, including sensitivity, specificity, positive predictive value (PPV), and negative predictive value (NPV).

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu Province Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No